CLINICAL TRIAL: NCT06640699
Title: The Effects of Neurophysiological Facilitation Techniques on Cardiopulmonary Parameters After Coronary Artery Bypass Graft Surgery
Brief Title: The Effects of Neurophysiological Facilitation Techniques After Coronary Artery Bypass Graft Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulOkanUnive
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Disease
Keywords: coronary artery bypass; respiratory function test; ventricular ejection fraction
MeSH Terms: conditions — Heart Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: participants will be blind to groups, outcomes assessor will be blind to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NFT Group (Experimental): NFT group will receive Phase I cardiac rehabilitation and neurophysiological facilitation techniques.
  Interventions: Other: exercise
- Control Group (Active Comparator): Control group will receive Phase I cardiac rehabilitation alone.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — exercises with using neurophysiological facilitation techniques and cardiac rehabilitation.

SUMMARY:
The aim of the study is to investigate the effects of neurophysiological facilitation techniques, applied in addition to Phase I cardiac rehabilitation in the early postoperative period after coronary artery bypass graft (CABG) surgery, on left ventricular function, respiratory functions, and functional capacity.

DETAILED DESCRIPTION:
In this prospective randomized controlled study, participants will be randomly divided into two groups: the control group, which will receive Phase I cardiac rehabilitation, and the treatment group, which will receive Phase I cardiac rehabilitation along with the application of neurophysiological facilitation techniques. The participants' left ventricular function, respiratory functions, and functional capacity will be assessed before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* First-time undergoing open-heart surgery
* Aged between 50 and 85 years
* Full cooperation

Exclusion Criteria:

* Presence of facial, sternum, or rib fractures
* Chronic renal failure
* Development of cerebrovascular events
* Cognitive function impairment
* Development of deep vein thrombosis in the postoperative period
* Presence of neuromuscular disease
* Presence of orthopedic disabilities
* Intubation duration longer than 24 hours
* Staying in intensive care for more than 48 hours

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ecocardiography device | 3 months
  ejection fraction will assess with ecocardiography.
spirometer | 3 months
  respiratory function test will assess with spirometer
6 Minutes walking test | 3 months
  functional capacity will assess with 6 minutes walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydın, PhD, Principal Investigator — Okan University

IPD SHARING:
Plan to Share IPD: No